CLINICAL TRIAL: NCT03563066
Title: Benralizumab Regulates Atopic Dermatitis Through Effects on Eosinophils, Basophils and Innate Lymphoid Type 2 Cells.
Brief Title: Effect of Benralizumab in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-16-12430
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2021-10

CONDITIONS: Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases
Keywords: Skin Lesions; Benralizumab; Eosinophils; Intra-dermal challenge; Anti-inflammatory agents; Physiological Effects of Drugs
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Benralizumab (Experimental): Fixed dose 30mg benralizumab.
  Interventions: Drug: Benralizumab
- Placebo Control (Placebo Comparator): Will appear identical in form to benralizumab arm.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Benralizumab — Subcutaneous benralizumab injections once per month for 3 months on Days 0, 28 & 56.
  Arms: Benralizumab
Drug: Placebo Control — Subcutaneous placebo injections once per month for 3 months on Days 0, 28 & 56.
  Arms: Placebo Control

SUMMARY:
Atopic Dermatitis (AD), also known as eczema, is a common skin disease characterized by itchy lesions. The prevalence of AD has increased over the past few decades, with 15-30% of children and 2-10%of adults being affected. The lesions of AD patients are very inflamed, with an increased number of inflammatory cells in the skin. There are not many medications available that are fully effective and can be used long-term for treatment of atopic dermatitis. Benralizumab is a monoclonal antibody used for treatment of a type of asthma called "eosinophilic asthma". Atopic dermatitis is also associated with elevated levels of eosinophils, and we would like to determine if benralizumab is effective in patients with atopic dermatitis. This is a randomized, double-blind, parallel group, placebo-controlled study will evaluate the effect of 3 doses of a fixed 30 mg dose of benralizumab administered subcutaneously (SC) every 4 weeks to patients with moderate-to-severe atopic dermatitis, on the severity of atopic dermatitis, and the cellular inflammation of skin lesions in these patients. Anti-inflammatory properties of benralizumab when a skin flare is induced in a controlled laboratory setting, in addition to the effects of benralizumab on skin that is already inflamed will be examined.It is hypothesized that benralizumab will attenuate eosinophilic inflammation in the skin.

DETAILED DESCRIPTION:
Patients with a history of moderate-to-severe atopic dermatitis will enter a screening period (Days -3 to -1) to assess responses to intradermal allergen challenge. Those developing a late cutaneous response 24 hours post-intradermal allergen challenge will be recruited for the study and have the size of the wheal/flare measured. A punch biopsy obtained from the challenge site and samples of peripheral blood and skin lesions will be obtained. Prior to randomization, skin lesions will be graded using the validated Eczema Area and Severity Index (EASI) Score as a baseline measure of the severity of disease. Patients will then be randomized 1:1 to benralizumab (30 mg SC monthly) or placebo, with dosing at days 0, 28 and 56 (± 3 days). On Day 64 (1 week after the last dose of study drug), an intradermal allergen challenge will be conducted to determine the effect of benralizumab on allergen-induced responses in skin. On Day 65 (24 hours post-intradermal allergen challenge), the size of the wheal/flare will be measured and a punch biopsy will be obtained from the challenge site and samples peripheral blood and skin lesions will be obtained. Skin lesions will be reassessed clinically on Day 65 using the EASI score to assess the effect of benralizumab on changes to the severity of disease. A safety followup visit will take place at week 20, which is 140 days after the first dose (12 weeks after the last dose/11 weeks after the last study procedure).

Primary endpoint

1. The number of eosinophils per millimetre squared of skin, measured 24 hours post intradermal allergen challenge, 65 days after the first dose. The number of eosinophils in the skin will be assessed by histological examination of a punch skin biopsy obtained from the site of the intradermal allergen challenge.

   Secondary endpoints
2. The size of the late cutaneous response, measured 24 hours post intradermal allergen challenge, 65 days after the first dose. The late cutaneous response will be calculated using the length and width of the wheal and flare response to a standardized amount of allergen extract.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 through 65 years of age.
2. Women of childbearing potential (WOCBP) must not be actively seeking pregnancy, and must use an effective form of birth control (confirmed by the Investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device (IUD)/ levonorgestrel Intrauterine system (IUS), Depo-Provera™ injections, oral contraceptive, and Evra Patch™ or Nuvaring™. WOCBP must agree to use effective method of birth control, as defined above, from enrolment, throughout the study duration and within 16 weeks after last dose of IP. They must demonstrate a negative serum pregnancy test at screening and demonstrate a negative urine pregnancy test immediately before each dose of study drug or placebo. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
   * Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
3. All male patients who are sexually active must agree to use an acceptable method of contraception (condom with or without spermicide, vasectomy) from the first dose of investigational product (IP) until 16 weeks after their last dose.
4. General good health
5. Moderate to severe atopic dermatitis
6. Able to understand and give written informed consent and has signed a written informed consent form approved by the investigator's Research Ethics Board (REB)

The following inclusion criteria must be met for entry into the dosing phase of the study:

1. Positive skin-prick test to common aeroallergens (including cat, dust mite, grass, pollen)
2. Positive late cutaneous response to intradermal allergen challenge

Exclusion Criteria:

1. History of anaphylaxis to any biologic therapy or vaccine
2. History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light headedness, as judged by the investigator
3. Any history or symptoms of cardiovascular disease, particularly coronary artery disease, arrhythmias, hypertension, or congestive heart failure
4. Any history or symptoms of significant neurologic disease, including transient ischemic attack (TIA), stroke, seizure disorder, or behavioral disturbances
5. Any history or symptoms of clinically significant autoimmune disease
6. Any history of clinically significant haematologic abnormality, including coagulopathy or any history of chronic treatment with anticoagulants (e.g. warfarin, etc) or antiplatelet agent (e.g, aspirin, etc)
7. Clinically significant abnormalities in laboratory test results at enrolment and during the screening period (including complete blood count, coagulation, chemistry panel and urinalysis) unless judged not significant by the investigator.
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.5 times the upper limit of normal (ULN) confirmed during screening period
9. Being pregnant or lactating or have positive serum pregnancy test at enrolment or positive urine pregnancy test during the study
10. Concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease
11. Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study
12. Presence of skin comorbidities that may interfere with study assessments
13. History of cancer: Patients who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent. Patients who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date of informed consent.
14. Patient who has a scheduled in-patient surgery or hospitalization during the study.
15. History of Guillain-Barré syndrome
16. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy
17. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Patients with a history of hepatitis B vaccination without history of hepatitis B are allowed to enrol
18. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test
19. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
20. Receipt of any marketed (eg omalizumab) or investigational biologic within 4 months or 5 half-lives prior to randomization is obtained, whichever is longer
21. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
22. Any allergen immunotherapy within 4 months prior to or throughout the study.
23. Having used any of the following treatments within 4 weeks before the Day -2 baseline visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during study:

    1. Immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon gamma (IFN-γ), Janus kinase inhibitors, azathioprine, methotrexate, etc.)
    2. Phototherapy for AD
24. Any cell-depleting agents including but not limited to rituximab: within 6 months before the baseline visit, or until lymphocyte count returns to normal, whichever is longer
25. Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (patients may continue using stable doses of such moisturizers if initiated before the screening visit)
26. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the baseline visit
27. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. Note: patients may be re-screened after infection resolves
28. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment
29. Planned or anticipated major surgical procedure during the patient's participation in this study
30. Receipt of live attenuated vaccines 30 days prior to the date of randomization. Receipt of inactive/killed vaccinations (eg, inactive influenza) are allowed provided they are not administered within 1 week before/after any IP administration.
31. Patient is a member of the investigational team or his/her immediate family
32. Pregnant woman
33. Previously received benralizumab (MEDI-563)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whetstone CE, Cusack RP, Price EL, Howie KJ, Stevens C, Al-Sajee D, Beaudin S, Wattie J, Alsaji N, Schlatman A, Luk V, O'Byrne PM, Inman MD, Sehmi R, Lima H, Gauvreau GM. Benralizumab Depletes IL-5Ralpha-Bearing Cells in Skin Lesions of Patients With Atopic Dermatitis. Clin Transl Allergy. 2025 Aug;15(8):e70090. doi: 10.1002/clt2.70090. PMID 40781582
- [Derived] Whetstone CE, Cusack RP, Price E, Howie K, Stevens C, Al-Sajee D, Beaudin S, Wattie J, Alsaji N, Schlatman A, Luk V, Ju X, O'Byrne P, Inman M, Sehmi R, Lima H, Gauvreau GM. Effect of benralizumab on inflammation in skin after intradermal allergen challenge in patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol Glob. 2024 Jul 22;3(4):100310. doi: 10.1016/j.jacig.2024.100310. eCollection 2024 Nov. PMID 39234416

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Benralizumab | Placebo Control
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total patients included in study
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo Control | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14) | 39 (14) | 40 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 9 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Allergen-induced Eosinophils in the Skin
Description: The primary objective is to evaluate the effect of benralizumab on the allergen-induced number of eosinophils in the skin assessed by histological examination compared to placebo. Intradermal saline challenge will be used as a control.
Time Frame: Day 65, 24 hours post-intradermal allergen challenge
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | Benralizumab | Placebo Control
Number analyzed (Participants) | 9 | 11
cells/mm2 | 11.95 (28.51) | 71.15 (130.1)

2. Secondary Outcome: Allergen-induced Late Phase Cutaneous Response
Description: To evaluate the effect of Benralizumab on the allergen-induced late phase cutaneous response by measuring the skin wheal compared to placebo.
Time Frame: Day 65, at 24 hours post-intradermal allergen challenge
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Benralizumab | Placebo Control
Number analyzed (Participants) | 9 | 11
millimeters | 18.89 (6.33) | 26.57 (12.07)

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Description: All AE and SAEs are reported.
Arm/Group | Benralizumab | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03563066/Prot_SAP_001.pdf